CLINICAL TRIAL: NCT02264483
Title: Assessment of the Degree of Pneumonia Underdiagnosis in Chronic Obstructive Pulmonary Disease (COPD) Exacerbations Using Chest Low-dose Computed Tomography (CT) and Comparison of Inflammatory Profile Between the Two Entities
Brief Title: Low-dose CT for Diagnosis of Pneumonia in COPD Exacerbations and Comparison of the Inflammatory Profile.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-EPO-2013-152
Record Dates: First submitted 2014-09-12; First posted 2014-10-15 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: COPD Exacerbation
Keywords: Pneumonia in COPD exacerbation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and sputum (supernatant)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD exacerbation: No intervention.
  The subjects will be divided in 2 subgroups according to the image study:
  * COPD exacerbation with pneumonia
  * COPD exacerbation without pneumonia
- COPD stable patients

SUMMARY:
* Hypothesis: There is an underdiagnosis of pneumonia in COPD (Chronic Obstructive Pulmonary Disease) exacerbations which could be demonstrated by performing low-dose chest CT. Differences in the inflammatory profile in sputum and blood in patients with and without pneumonia can be seen.

* Objective: To assess the degree of underdiagnosis of pneumonia in COPD exacerbations, using chest low-dose CT and to compare clinical and inflammatory differences in blood and sputum between patients with and without pneumonia.

*Material and Methods: Prospective observational study including 75 patients with the diagnosis of COPD at the time of an exacerbation and with criteria for a respiratory tract infection. At the time of inclusion clinical features, blood and sputum analysis, chest X-ray and chest low-dose CT are performed. The investigators divide the patients into two groups according to the existence of pneumonia and the inflammatory pattern in blood (inflammatory markers) and sputum (cell populations and inflammatory markers) is compared between the two branches.

ELIGIBILITY:
INCLUSION CRITERIA

* clinical and spirometric diagnosis of COPD.
* for study group: clinical symptoms of exacerbation and infection of low airway.
* Signed informed consent.

EXCLUSION CRITERIA

* No acceptance of informed consent.
* The STUDY GROUP: treatment with antibiotic more tan 2 days before consultation.
* Another entity known pulmonology other than COPD (non-obstructive disorders, bronchiectasis, interstitial lung disease patients, severe pulmonary hypertension, hypoventilation).
* Chronic treatment with oral corticosteroids or immunosuppressive drug.
* severe organ comorbidity such as cancer in advanced or terminal phase, pulmonary tuberculosis with important involvement, severe pneumoconiosis.
* Severe alteration of nutritional status.
* Heart disease evolved.
* Limitation for understanding the study (including psychiatric disorder, language problem, social or cultural differences, etc.).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients with an exacerbation of their disease and symptoms of respiratory infection, wich come to visit at outpatient pneumologic clinic.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with an exacerbation of their disease who have a Pneumonia diagnosed by low dose - CT (not detected by chest X-Ray). | 1 year and a half

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Solanes, MD PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain